CLINICAL TRIAL: NCT02270879
Title: Multi-formula Optimization of Second Eye Refinement According to Direction of the Prediction Error of the First Eye
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Baixo Vouga (Other)
Responsible Party: Principal Investigator, Pedro Gil, MD, MSc, Centro Hospitalar do Baixo Vouga
Other Study IDs: CHBaixoVouga
Record Dates: First submitted 2014-10-18; First posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Main group: Patients having performed bilateral consecutive cataract surgery between 1st October 2012 and 24th April 2014 in a single ophthalmological center (Centro Hospitalar Baixo Vouga, Portugal).
  Interventions: Procedure: Phacoemulsification cataract surgery

INTERVENTIONS:
Procedure: Phacoemulsification cataract surgery — Phacoemulsification of cataract (opacified lens) using clear corneal approach. Implantation of a intra-ocular lens in the capsular bag

SUMMARY:
Prediction errors for the first (PE1) and second eyes (PE2) were obtained in the intra-ocular lens power calculation for 4 formulae (HofferQ, SRK II, SRK/T and Holladay 1). The optimal correction factor for each formula was determined as the one resulting in the lowest mean absolute error. A similar analysis was performed in the negative and positive PE1 subgroups.

DETAILED DESCRIPTION:
Retrospective case series study. A retrospective chart review was conducted, which included demographics (age and gender) and several parameters for both the first and second eyes: surgery date, axial length, keratometric corneal power in 2 meridians, predicted intra-ocular lens (IOL) power recommended for plano target in each formulae (HofferQ, SRK II, SRK/T and Holladay 1), implanted IOL power, predicted post-operative refraction for the implanted IOL for the 4 formulae, observed post-operative refraction in spherical equivalent and post-operative best corrected visual acuity. The prediction error was calculated for the first eye (PE1) as the difference between the observed post-operative refraction in spherical equivalent and the predicted post-operative refraction by the IOL Master for the implanted IOL. This was obtained for the 4 formulae. The prediction error for the second eye (PE2) was obtained in a similar fashion. The optimal partial adjustment for second eye refinement was obtained subtracting a portion of the PE1 from the PE2 (PE2-xPE1, where 0≤x≤1) for the 4 formulae. The optimal correction factor was determined for all formulae by using an array of different proportions of PE1 that were applied to the second eye. The values ranged from 10% to 100%, with increments of 10% each.

ELIGIBILITY:
Inclusion Criteria:

* Patients having performed bilateral cataract surgery between 1st October 2012 and 24th April 2014 in a single ophthalmological center (Centro Hospitalar Baixo Vouga, Portugal)

Exclusion Criteria:

* Inadequate follow-up
* Incomplete medical records
* Previous or combined ocular surgery
* Manual extracapsular cataract extraction and not phacoemulsification
* Corneal sutures
* Implantation of any other IOL type different from Abbott Tecnis® 1-piece IOL (Abbott Laboratories Inc., Illinois, USA), ZCB00
* IOL implanted in the sulcus
* Intra or postoperative complication
* Post-operative best corrected visual acuity worse than 5/10
* Corneal astigmatism>3.00 D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a single ophthalmological center (Centro Hospitalar Baixo Vouga, Portugal) admitted for bilateral consecutive cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Second eye mean absolute error (mean of the absolute value of the prediction error) | 6 weeks after date of cataract surgery

SECONDARY OUTCOMES:
Percentage of second eyes with a post-operative refraction within ±0.50 D and ±1.00 D of the targeted refraction | 6 weeks after date of cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gil, MD, MSc, Principal Investigator — Centro Hospitalar do Baixo Vouga